CLINICAL TRIAL: NCT02831049
Title: Effects of a New Behavioral Intervention on Alcohol Craving and Drinking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 999916140; 16-DA-N140
Record Dates: First submitted 2016-07-09; First posted 2016-07-13 (Estimated); Results first posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-10-09

CONDITIONS: Alcohol Drinking; Alcohol Drinking Related Problems
Keywords: Reconsolidation
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group: Alcohol retrieval / Alcohol extinction (A/A) (Experimental): Participant drinks an alcoholic beverage (individualized to produce a 0.06 g/dL blood alcohol content). Participant is then repeatedly presented with alcohol-associated cues without further drinking. Participant completes four sessions of memory retrieval and extinction portions, a novel behavioral procedure for reduction of craving and drinking, in problem drinkers.
  Interventions: Behavioral: Retrieval-extinction; Behavioral: Alcohol-related cues
- Control Group A: Soft-drink retrieval / Alcohol extinction (S/A) (Active Comparator): Participant undergoes retrieval with with soft drink cues followed by extinction with alcohol-related cues without further drinking. Participant completes four sessions of memory retrieval and extinction portions, a novel behavioral procedure for reduction of craving and drinking, in problem drinkers.
  Interventions: Behavioral: Retrieval-extinction; Behavioral: Alcohol-related cues
- Control Group B: Alcohol retrieval / Soft-drink extinction (A/S) (Active Comparator): Participant drinks an alcoholic beverage (individualized to produce a 0.06 g/dL blood alcohol content). Participant is then repeatedly presented with soft drink-associated cues without further drinking. Participant completes four sessions of memory retrieval and extinction portions, a novel behavioral procedure for reduction of craving and drinking, in problem drinkers.
  Interventions: Behavioral: Retrieval-extinction; Behavioral: Soft-drink related cues

INTERVENTIONS:
Behavioral: Retrieval-extinction — Memory retrieval-extinction is a novel behavioral procedure for reduction of craving and drinking in problem drinkers.
Behavioral: Alcohol-related cues — Alcohol related cues
  Arms: Control Group A: Soft-drink retrieval / Alcohol extinction (S/A); Experimental Group: Alcohol retrieval / Alcohol extinction (A/A)
Behavioral: Soft-drink related cues — Soft drink related cues
  Arms: Control Group B: Alcohol retrieval / Soft-drink extinction (A/S)

SUMMARY:
Background:

Sights, sounds, and smells can be associated with alcohol and tempt people to drink. The connection between encountering cues and wanting to drink might be reduced by behavioral techniques, like giving the cues at certain times, in certain circumstances.

Objective:

To see if visual imagery and behavioral techniques can reduce alcohol craving and drinking.

Eligibility:

Healthy people ages 21 to 65 years old who are mildly concerned about their drinking and have had these habits in the past 3 months:

* Women: More than three (3) drinks any single day or more than seven (7) drinks per week
* Men: More than four (4) drinks any single day or more than 14 drinks per week

Design:

* Participants will be screened with medical history, physical exam, blood tests, alcohol breath tests, hepatitis tests, and alcohol and drug use questionnaires.
* Participants will get a smartphone to carry throughout the study. They will use it to report on their drinking, moods, and activities daily. The phone's global positioning system (GPS) will record their locations throughout each day.
* There will be six (6) study visits approximately over four (4) weeks. Visits will last up to four (4) hours, but the final visit may last up to seven (7) hours. Visits include the following:

  * Not drinking alcohol or using illicit or over-the-counter drugs at least 24 hours before each visit
  * Providing urine and breath samples.
  * Exposure to various cues: Participants' reactions will be monitored by measuring heart rate, blood pressure, and skin temperature.
  * Drinking alcohol or soft drinks: For visits with alcohol, transportation to and from the visit will be provided.
* About a month after the last visit, participants will be called to ask about their drinking and cravings.

DETAILED DESCRIPTION:
Objective: To evaluate alcohol memory retrieval-extinction, a novel behavioral procedure for reduction of craving and drinking, in problem drinkers.

Study population: We will collect evaluable data from up to 75 participants. Participants are evaluable if they complete ecological momentary assessment (EMA, described below). All participants will be adult alcohol drinkers (men: > 14 drinks/week or > 4 drinks/day; women: > 7 drinks/week or > 3 drinks/day) whose drinking scores as hazardous on the Alcohol Use Disorders Identification Test. Participants will not be seeking treatment for an alcohol-use disorder, be physiologically dependent on alcohol, or have other drug use disorders. Participants can have nicotine use disorder.

Design: A randomized study with three groups. Participants will use smartphones to provide geotagged reports of alcohol craving and drinking in daily life (EMA reports) before, between, and after a series of laboratory sessions. During sessions, participants will drink an alcoholic beverage (individualized to produce a 0.06 g/dL blood alcohol content) or a soft drink. Participants will then be repeatedly presented with alcohol or soft drink-associated cues without further drinking. These are the memory retrieval and extinction portions, respectively, of memory retrieval-extinction. Previous studies suggest this procedure can robustly reduce Pavlovian associations between cues and responses such as craving. The mechanism seems to involve memory reconsolidation, in which freshly retrieved associations (e.g. drink cues and consumption - pleasant effects) become more vulnerable to disruption by extinction.

Three groups will be tested: (1) alcohol retrieval / alcohol extinction will be compared to (2) soft-drink retrieval / alcohol extinction and (3) alcohol retrieval / soft-drink extinction. Before and after retrieval-extinction, participants will be tested for alcohol craving and cue-induced physiological responses in laboratory sessions. Retrieval-extinction will be followed by approximately one week of follow-up EMA reporting, with telephone contact approximately 30 days thereafter.

Outcome parameters:

* The co-primary outcome measures are: self-reported alcohol craving in the laboratory sessions before and after retrieval-extinction, and EMA reports of alcohol craving and drinking. Daily-life responses are important because the version of retrieval-extinction we will be using, with retrieval induced by drinking alcohol itself, rather than alcohol cues alone, may be especially likely to have effects that generalize from the laboratory to daily life.
* Secondary outcome measures are: self-reported alcohol craving and drinking at 30-day follow-up

ELIGIBILITY:
INCLUSION CRITERIA:

* Age between 21 and 65 years inclusive
* Drinking at high levels for at least 10 different weeks during the last 90 days. High-level drinking for a given week can be either of the following:

  * For women, more than 3 drinks on any single day that week, or more than 7 drinks that week
  * For men, more than 4 drinks on any single day that week, or more than 14 drinks that week
* A score greater than or equal to 8 and less than or equal to 15 on the self-report version of the Alcohol Use Disorders Identification Test (AUDIT), with endorsement of at least one item other than 1-3, because 1-3 assess only consumption, not concern or consequences
* Self-report of liking or having neutral feelings about the sight and smell of alcoholic beverages
* For women,

  * practicing an effective method of birth control before entry and throughout the study (or postmenopausal for at least one year, or surgically sterile)
  * negative urine pregnancy test at each visit.
  * Effective methods of birth control are those approved by the Food and Drug Administration (FDA) used as described in the FDA Birth Control Guide These methods are: (1) intrauterine device (IUD) copper; (2) IUD with progestin; (3) implantable rod; (4) contraceptive shot/injection; (5) oral contraceptives (combined pill, progestin-only pill, or extended/continuous-use combined pill); (6) contraceptive patch; (7) vaginal contraceptive ring; (8) diaphragm with spermicide; (9) sponge with spermicide; (10) cervical cap with spermicide; (11) male condom; (12) female condom; (13) male partner with a vasectomy. Abstinence from sexual intercourse is also an effective method of birth control.

EXCLUSION CRITERIA:

* Risk of alcohol withdrawal, as determined by any of the following:

  * a score less than 8 or greater than 15 on the Clinical Institute Withdrawal Assessment for Alcohol, Revised (CIWA-Ar) following a negative breath test for alcohol (i.e., blood alcohol concentration of 0.0)
  * lifetime history of delirium tremens or seizures (related to alcohol or not),
  * endorsement of a drinking to avoid withdrawal symptom on the Structured Clinical Interview for Diagnostic and Statistical Manual Disorders (SCID) or Mini International Neuropsychiatric Interview (M.I.N.I) (M.I.N.I. Section I, Alcohol Use Disorder, items k1 and/or k2 answered affirmatively with counselor's evaluation to verify that symptoms indicated in item k1 are related to the individual's cutting down on drinking and/or the response to item k2 refers to withdrawal symptoms and not hangover);
  * OR physician's judgment.
* Currently trying to quit drinking, or planning to quit or reduce alcohol drinking via formal treatment or support-group attendance in the next six months;
* For women: pregnancy, breastfeeding, or planning to become pregnant during the experiment
* Current liver disease or dysfunction, assessed by physical examination and medical history; and hepatitis C, chronic hepatitis B, or other current liver disease or dysfunction as assessed by physical examination and medical history or as reflected in blood levels more than 5 times the upper limit of normal in any of the following: aspartate transaminase (AST), alanine transaminase (ALT), or gamma-glutamyltransferase (GGT)
* Any other medical illness or condition that in the judgment of the investigators is incompatible with alcohol consumption
* Current use of prescription or over-the-counter medications or herbal products for which drinking alcohol is strictly prohibited. When the metabolic half-life of the medication/product is known, we will require at least 7 half-lives to have elapsed before any session involving alcohol consumption. If the half-life is not known (as might be the case for some herbal preparations), we will require at least 7 days to have elapsed since the last use before any session involving alcohol consumption
* Substance-use disorder for any drug(s) other than alcohol or nicotine in the previous 12 months
* Past or present diagnosis of bipolar disorder or any psychotic disorder; any history of suicide attempt or current suicidal ideation; present diagnosis of uncontrolled or untreated mood or anxiety disorder
* Cognitive impairment severe enough to preclude informed consent or valid self-report

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2020-04-21 (Actual); Study Completion 2020-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H Epstein, M.D, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Some health information collected may be placed into one or more scientific databases after it has been stripped of identifiers such as name, address or account number, so that it may be used for future research on any topic and shared broadly for research purposes. A researcher who wants to study the information must apply to the database and be approved.
Access Criteria: We will share some protocol data with our scientific research partners inside or outside the NIH. Research partners outside the NIH sign an agreement with the NIH to share data. This agreement indicates the type of data that can be shared and what can be done with those data.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Group: Alcohol Retrieval / Alcohol Extinction (A/A) | Control Group A: Soft-drink Retrieval / Alcohol Extinction (S/A) | Control Group B: Alcohol Retrieval / Soft-drink Extinction (A/S)
Started | 7 | 8 | 8
Completed | 6 | 7 | 6
Not Completed | 1 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Pandemic shutdown | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group: Alcohol Retrieval / Alcohol Extinction (A/A) | Control Group A: Soft-drink Retrieval / Alcohol Extinction (S/A) | Control Group B: Alcohol Retrieval / Soft-drink Extinction (A/S) | Total
Number analyzed (Participants) | 7 | 8 | 8 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 8 | 23
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 9
  Male | 4 | 5 | 5 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 6 | 8 | 7 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 4 | 4 | 8
  White | 6 | 2 | 4 | 12
  More than one race | 0 | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 8 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in Self-reported Alcohol Craving in the Laboratory Sessions
Description: Participants were presented with alcohol cues and an alcohol-containing beverage in the laboratory sessions then cue-elicited craving was measured on a visual analogue scale using the question, "How much do want a drink right now?" on a scale of 0 = "I don't want a drink at all," to 100 = "I really want a drink". Higher score indicates more alcohol craving.
  The procedure was done in four intervention sessions, called retrieval-extinction sessions, and then in a test session as follows: Tests of renewal (control context was extinction context; challenge context was novel context) and reinstatement (by a priming dose of alcohol) were used to assess the success of the retrieval-extinction intervention. The outcome measure in the final session was changes in craving before versus after renewal, and again after reinstatement.
  Results are expressed as the estimated mean change in scores (after cues minus before cues).
Time Frame: Up to 75 minutes during trial sessions
Population: All participants who completed the study
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Experimental Group: Alcohol Retrieval / Alcohol Extinction (A/A) | Control Group A: Soft-drink Retrieval / Alcohol Extinction (S/A) | Control Group B: Alcohol Retrieval / Soft-drink Extinction (A/S)
Number analyzed (Participants) | 6 | 7 | 6
units on a scale
  Extinction context | 11.7 [-1.3 to 24.0] | 20.1 [6.9 to 33.0] | 15.3 [1.1 to 29.1]
  Novel context | 10.0 [-3.4 to 23.4] | 33.7 [19.4 to 48.2] | 16.1 [1.7 to 30.5]

2. Primary Outcome: Self-reported Alcohol Craving in the Laboratory Sessions - Reinstatement Trial
Description: Participants were presented with soft drink to drink, then craving was measured. Next participants were presented with alcohol to drink followed by craving measurement. Cue-elicited craving was measured on a visual analogue scale using the question, "How much do want a drink right now?" on a scale of 0 = "I don't want a drink at all," to 100 = "I really want a drink". Higher score indicates more alcohol craving.
  This outcome used a reinstatement procedure in which, instead of alcohol-related cues, the unconditioned stimulus (alcohol) is presented (participants are provided with an alcoholic beverage), to determine whether the extinguished response (craving) reappears (a "priming" effect).
  Results are expressed as the estimated mean change scores (after cues minus before cues).
Time Frame: Up to 90 minutes during reinstatement trials in a single day visit
Population: All participants who completed the study.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Experimental Group: Alcohol Retrieval / Alcohol Extinction (A/A) | Control Group A: Soft-drink Retrieval / Alcohol Extinction (S/A) | Control Group B: Alcohol Retrieval / Soft-drink Extinction (A/S)
Number analyzed (Participants) | 6 | 7 | 6
units on a scale | 18.7 [11.6 to 28.3] | 24.7 [17.7 to 34.1] | 9.7 [5.7 to 16.4]

3. Primary Outcome: Drinking in Daily Life Assessed With the Ecological Momentary Assessment (EMA)
Description: Participants drinking over the course of the study was assessed through ecological momentary assessment (EMA), based on self-reports provided through random-prompt and event-contingent entries. Participants reported drinking or not report drinking on each day. EMA uses real-time assessments of behavior and emotion on mobile electronic devices.
  Results are expressed as the estimated probability of reporting drinking within a day.
Time Frame: 22-37 days
Population: All participants who completed the study
Measure: Mean (95% Confidence Interval); unit: Probability of reported drinking/day
Arm/Group | Experimental Group: Alcohol Retrieval / Alcohol Extinction (A/A) | Control Group A: Soft-drink Retrieval / Alcohol Extinction (S/A) | Control Group B: Alcohol Retrieval / Soft-drink Extinction (A/S)
Number analyzed (Participants) | 6 | 7 | 6
Probability of reported drinking/day | 0.799 [0.616 to 0.906] | 0.549 [0.353 to 0.729] | 0.513 [0.285 to 0.733]

4. Primary Outcome: Craving in Daily Life Assessed With Event-contingent Ecological Momentary Assessment (EMA)
Description: Participants craving over the course of the study was assessed through ecological momentary assessment (EMA), based on self-reports provided through event-contingent entries initiated by the participant whenever they feel a craving, urge, or temptation to drink, in response to the question on a visual analogue scale, "How much do want a drink right now?" on a scale of 0 = "I don't want a drink at all," to 100 = "I really want a drink". Higher score indicates more alcohol craving.
  Results are expressed as the estimated mean of level of craving
Time Frame: 22-37 days
Population: All participants who completed the study.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Experimental Group: Alcohol Retrieval / Alcohol Extinction (A/A) | Control Group A: Soft-drink Retrieval / Alcohol Extinction (S/A) | Control Group B: Alcohol Retrieval / Soft-drink Extinction (A/S)
Number analyzed (Participants) | 6 | 7 | 6
units on a scale | 5.5 [0.8 to 20.6] | 7.1 [1.6 to 22.7] | 13.8 [3.5 to 40.2]

5. Primary Outcome: Craving in Daily Life Assessed With Random-prompt Ecological Momentary Assessment (EMA)
Description: Participant craving over the course of the study was assessed through ecological momentary assessment , based on self-reports provided through random-prompt entries in response to the question on a visual analogue scale, "How much do want a drink right now?" on a scale of 0 = "I don't want a drink at all," to 100 = "I really want a drink". Higher score indicates more alcohol craving.
  Results are expressed as the estimated mean of level of craving.
Time Frame: 22-37 days
Population: All participants who completed the study.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Experimental Group: Alcohol Retrieval / Alcohol Extinction (A/A) | Control Group A: Soft-drink Retrieval / Alcohol Extinction (S/A) | Control Group B: Alcohol Retrieval / Soft-drink Extinction (A/S)
Number analyzed (Participants) | 6 | 7 | 6
units on a scale | 24.8 [7.8 to 55.0] | 28.1 [10.2 to 55.7] | 7.2 [1.4 to 23.2]

6. Secondary Outcome: Change in Alcohol Craving Assessed Using the Penn Alcohol Craving Scale
Description: Penn Alcohol Craving Scale (PACS) is a self-reported measure that inquires about the frequency, intensity, and duration of craving, the ability to resist drinking, and overall rating of craving for alcohol on a week's timescale, providing a retrospective measure of craving. PACS is a five item questionnaire with each item scored from 0 to 6. Total score range from 0 to 30. Higher score indicates more frequent craving.
  Craving was measured in once on the first day of treatment and again in a phone call 30 days after last laboratory session.
  Outcome was analyzed as the change in score (day 30 score minus day 1 score).
Time Frame: Day 1 of study and 30 days after the final laboratory session
Population: All participants who completed the study.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Experimental Group: Alcohol Retrieval / Alcohol Extinction (A/A) | Control Group A: Soft-drink Retrieval / Alcohol Extinction (S/A) | Control Group B: Alcohol Retrieval / Soft-drink Extinction (A/S)
Number analyzed (Participants) | 6 | 7 | 6
units on a scale | -0.3 [-4.1 to 3.5] | 0.4 [-3.1 to 3.9] | 1.6 [-2.6 to 5.7]

ADVERSE EVENTS:
Time Frame: Up to 3 months from start of study
Arm/Group | Experimental Group: Alcohol Retrieval / Alcohol Extinction (A/A) | Control Group A: Soft-drink Retrieval / Alcohol Extinction (S/A) | Control Group B: Alcohol Retrieval / Soft-drink Extinction (A/S)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/7 | 1/8 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Group: Alcohol Retrieval / Alcohol Extinction (A/A) (N=7) | Control Group A: Soft-drink Retrieval / Alcohol Extinction (S/A) (N=8) | Control Group B: Alcohol Retrieval / Soft-drink Extinction (A/S) (N=8)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Menstrual discomfort (Reproductive system and breast disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/49/NCT02831049/Prot_SAP_000.pdf